CLINICAL TRIAL: NCT05578469
Title: Effect of Different Surgical Treatment of Marfan Syndrome With Subluxation Lens
Brief Title: Surgical Treatment of Marfan Syndrome With Subluxation Lens
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0765
Record Dates: First submitted 2022-10-11; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-09

CONDITIONS: Marfan Syndrome; Lens Subluxation or Dislocation
MeSH Terms: conditions — Marfan Syndrome; Lens Subluxation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- posterior chamber intraocular lens(IOL) implantation with a Cionni capsular tension ring (CTR)
  Interventions: Procedure: surgical treatment of Marfan Syndrome with subluxation lens
- sutured scleral fixation of posterior chamber IOL/ posterior chamber IOL and CTR
  Interventions: Procedure: surgical treatment of Marfan Syndrome with subluxation lens

INTERVENTIONS:
Procedure: surgical treatment of Marfan Syndrome with subluxation lens — different surgical treatment of Marfan Syndrome with subluxation lens

SUMMARY:
To analyze the postoperative visual effects, and to compare the safety and efficacy of different surgical treatment with of Marfan Syndrome with subluxation lens.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with MFS according to the revised Ghent etiology.
2. refractive errors difficult to correct.
3. pupillary block glaucoma caused by severe dislocation of the lens

Exclusion Criteria:

Keratoconus, late glaucoma, uveitis, history of traumatic lens dislocation, and preoperative retinal rupture with or without retinal detachment (RD)

Ages: 8 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with lens dislocation of Marfan syndrome who accepted different surgical treatments
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Uncorrected distance visual acuity | 1 month postoperatively
Uncorrected distance visual acuity | 3 month postoperatively
Corrected distance visual acuity | 1 month postoperatively
Corrected distance visual acuity | 3 month postoperatively
intraocular pressure | 1 month postoperatively
intraocular pressure | 3 month postoperatively
postoperative complication | Early and late stages

SECONDARY OUTCOMES:
Postoperative astigmatism and astigmatism axial of cornea | 1 month postoperatively
Postoperative astigmatism and astigmatism axial of cornea | 3 month postoperatively
endothelial cell count | 1 month postoperatively
endothelial cell count | 3 month postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No